CLINICAL TRIAL: NCT01484405
Title: Anterolateral Versus Posterior Approach for Total Hip Arthroplasty After Displaced Femoral Neck Fracture
Acronym: THA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment.
Sponsor: Florida Orthopaedic Institute (Network)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THA
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Femur Fracture
Keywords: surgical approach for total hip arthroplasty
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- anterolateral approach (Other): surgical intervention THA anterolateral approach
  Interventions: Procedure: anterolateral approach
- posterior approach (Other): surgical intervention THA posterior approach
  Interventions: Procedure: posterior approach

INTERVENTIONS:
Procedure: posterior approach — Surgical approach for Total Hip Arthroplasty
  Other Names: Total hip Athroplasty following fracture
  Arms: posterior approach
Procedure: anterolateral approach — anterolateral surgical approach
  Other Names: Total hip Athroplasty following fracture
  Arms: anterolateral approach

SUMMARY:
There are two surgical approaches (incision types) used by surgeons who do total hip replacements. The purpose of this study is to determine which type of surgical approach (incision type) produces the best results for patients who have a total hip replacement.

Null Hypothesis : There is no difference in complication rate, functional outcome, surgical time, or blood loss when comparing outcomes in patients receiving THA to hemiarthroplasty or ORIF for femoral neck fractures.

DETAILED DESCRIPTION:
Patients undergoing Total hip Arthroplasty following displaced femoral neck fracture, will be consented and randomized to one of two surgical approaches ( anterior or posterior).

ELIGIBILITY:
Inclusion Criteria:

* Displaced femoral neck fracture
* Age 65 years or older
* Acute, femoral neck fracture

Exclusion Criteria:

Cognitive impairment

* Active Infection
* Limited functional capacity (nursing home resident, non-ambulatory, severe cardiorespiratory disease)
* Limited life expectancy
* Pathologic fracture (tumor)
* Acetabular fractures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
dislocation rates | 12 months
  Radiographic variables: AP and lateral views of hip and pelvis

SECONDARY OUTCOMES:
other complications | 12 months
  Hospital readmission, reoperation

CONTACTS AND LOCATIONS:
Overall Officials: David Watson, MD, Principal Investigator — Florida Orthopaedic Institute
Locations (2):
- United States (2):
  - Tampa general Hospital, Tampa, Florida
  - St Josephs Hospital, Tampa, Florida